CLINICAL TRIAL: NCT07062224
Title: Impact of a Probiotic Supplement on Gut Microbiota and Glycemic Control in Patients With Type 1 Diabetes Mellitus: A Randomized Double-Blind Clinical Trial
Brief Title: Effect of a Probiotic Supplement on Gut Microbiota and Glycemic Control in Patients With Type 1 Diabetes (PRODIAB)
Acronym: PRODIAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Mª Teresa Mercader Ros, Principal Investigator and Academic Secretary of the Bachelor's Degree in Human Nutrition and Dietetics at UCAM, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE122401
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Diabete Type 1
Keywords: Gut microbiota; Probiotic supplement; Zonulin; Calprotectin; Type 1 Diabetes; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This is a 2x2 factorial, randomized, double-blind clinical trial including adults with type 1 diabetes and healthy controls. Participants in both groups will be randomly assigned to receive either a probiotic/prebiotic supplement or a placebo. The intervention period will last approximately 98 days. The design allows for the evaluation of the independent and combined effects of participant type (T1D vs. healthy) and intervention (supplement vs. placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. Participants, investigators, care providers, and outcomes assessors are unaware of the group assignments. The probiotic and placebo supplements are identical in appearance and packaging, and group codes will remain confidential until after data analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Type 1 Diabetes - Supplement (Experimental): Participants with type 1 diabetes mellitus will receive a daily 10 mL gel supplement containing 4000 mg of inulin and 1000 mg of tyndallized probiotics for approximately 98 days. The supplement is designed to modulate gut microbiota and improve glycemic control.
  Interventions: Dietary Supplement: Probiotic/Prebiotic Supplement
- Type 1 Diabetes - Placebo (Experimental): Participants with type 1 diabetes mellitus will receive a daily 10 mL placebo gel without active ingredients for approximately 98 days. The placebo is organoleptically identical to the supplement to maintain blinding.
  Interventions: Dietary Supplement: Placebo Gel
- Healthy Controls - Supplement (Experimental): Healthy participants will receive a daily 10 mL gel supplement containing 4000 mg of inulin and 1000 mg of tyndallized probiotics for approximately 98 days. This arm allows comparison of microbiota and metabolic responses between diabetic and non-diabetic individuals.
  Interventions: Dietary Supplement: Probiotic/Prebiotic Supplement
- Healthy Controls - Placebo (Experimental): Healthy participants will receive a daily 10 mL placebo gel without active ingredients for approximately 98 days. The placebo is identical in appearance and flavor to the active supplement.
  Interventions: Dietary Supplement: Placebo Gel

INTERVENTIONS:
Dietary Supplement: Probiotic/Prebiotic Supplement — Oral dietary supplement in gel form (10 mL per day) containing 4000 mg of inulin and 1000 mg of tyndallized probiotics. Administered once daily for approximately 98 consecutive days. Produced by Martínez Nieto S.A. (MARNYS®). Intended to modulate gut microbiota and improve glycemic and inflammatory markers.
  Arms: Healthy Controls - Supplement; Type 1 Diabetes - Supplement
Dietary Supplement: Placebo Gel — Oral placebo in gel form (10 mL per day), identical in appearance, texture, and taste to the active supplement, but without probiotic or prebiotic components. Administered once daily for 98 days to maintain blinding and control effects.
  Arms: Healthy Controls - Placebo; Type 1 Diabetes - Placebo

SUMMARY:
This randomized, double-blind clinical trial aims to evaluate the effect of a probiotic supplement on gut microbiota composition and glycemic control in adults with type 1 diabetes mellitus. A secondary comparison will be made with a healthy control group. Participants will be assigned to receive either a probiotic or a placebo for 98 days. Stool samples and metabolic parameters will be collected at baseline and after the intervention period. The study seeks to better understand how modulation of the intestinal microbiota may influence glucose regulation in people with type 1 diabetes.

DETAILED DESCRIPTION:
This randomized, double-blind clinical trial aims to evaluate the impact of a nutritional supplement composed of inulin (prebiotic) and tyndallized probiotics (paraprobiotics) on gut microbiota composition, intestinal barrier integrity, and glycemic control in individuals with type 1 diabetes mellitus (T1D). A total of 80 participants will be recruited: 40 with T1D and 40 healthy controls. Each group will be randomly assigned to receive either the active supplement or a placebo for a period of approximately 98 days.

The study will include pre- and post-intervention assessments using stool samples (for microbiota analysis and intestinal inflammation markers like zonulin and calprotectin), continuous glucose monitor (CGM) data, blood tests (for glycemic, hepatic, renal, and lipid profiles), body composition analysis by bioimpedance (including phase angle), and validated questionnaires assessing gastrointestinal symptoms, lifestyle, dietary intake, and diabetes-related quality of life.

The main objectives are to analyze changes in gut microbiota diversity and composition, assess effects on intestinal permeability and inflammation, evaluate the safety and tolerability of the supplement, and determine its impact on metabolic markers such as fasting glucose, HbA1c, glycemic variability, and HOMA-IR.

This project seeks to explore microbiota modulation as a potential complementary therapeutic strategy for improving glycemic control and metabolic health in individuals with T1D. The supplement will be provided in 10 mL gel sticks, containing 4000 mg of inulin and 1000 mg of tyndallized probiotics, taken once daily. The intervention period has been strategically planned to avoid holidays and vacation times to ensure adherence and minimize lifestyle variability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Ability to understand and sign the informed consent form.
* For the patient group: diagnosis of type 1 diabetes with at least 1 year of disease progression.
* For the control group: healthy individuals without a diagnosis of diabetes or other metabolic disorders.
* No use of antibiotics, probiotics, or prebiotics during the 4 weeks prior to the study start.
* Willingness to comply with the study protocol and attend scheduled visits.

Exclusion Criteria:

* Current use of probiotics, prebiotics, or antibiotics.
* Chronic gastrointestinal diseases (e.g., inflammatory bowel disease, irritable bowel syndrome).
* Pregnancy or breastfeeding.
* Participation in another clinical trial within the past 3 months.
* Immunosuppressive diseases, active cancer, or treatment with immunosuppressants.
* Known allergy or intolerance to any component of the supplement or placebo.
* Excessive alcohol or drug use.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in gut microbiota composition | Baseline and 98 days post-intervention
  Variation in the relative abundance and diversity of gut microbiota species assessed by 16S rRNA sequencing from stool samples collected at baseline and after 98 days of intervention.

SECONDARY OUTCOMES:
Change in fasting glucose [Time Frame: Day 1 and Day 98] | Baseline and 98 days post-intervention
  Assessment of changes in fasting glucose levels (mg/dL) via blood test.
Change in HbA1c [Time Frame: Day 1 and Day 98] | Baseline and 98 days post-intervention
  Assessment of changes in glycated hemoglobin levels (HbA1c, %) via blood test.
Change in fasting insulin [Time Frame: Day 1 and Day 98] | Baseline and 98 days post-intervention
  Assessment of changes in fasting insulin levels via blood test. μU/mL
Change in HOMA-IR index [Time Frame: Day 1 and Day 98] | Baseline and 98 days post-intervention
  Assessment of changes in insulin resistance estimated using the HOMA-IR index.
Change in time in range (70-180 mg/dL) [Time Frame: 3 months] | Baseline and 98 days post-intervention
  Assessment of the percentage of time that glucose levels are within the target range using continuous glucose monitoring (CGM).
Change in time above range (>180 mg/dL) [Time Frame: 3 months] | Baseline and 98 days post-intervention
  Assessment of the percentage of time with hyperglycemia using CGM.
Change in time below range (<70 mg/dL) [Time Frame: 3 months] | Baseline and 98 days post-intervention
  Assessment of the percentage of time with hypoglycemia using CGM.
Change in mean glucose [Time Frame: 3 months] | Baseline and 98 days post-intervention
  Assessment of average glucose concentration (mg/dL) using CGM.
Change in glucose variability [Time Frame: 3 months] | Baseline and 98 days post-intervention
  Assessment of glucose coefficient of variation (%) using CGM.
Change in plasma zonulin levels [Time Frame: Day 1 and Day 98] | Baseline and 98 days post-intervention
  Zonulin levels will be measured in fasting plasma samples using ELISA at baseline and after the intervention (ng/mL).
Change in fecal calprotectin levels [Time Frame: Day 1 and Day 98] | Baseline and 98 days post-intervention
  Calprotectin levels will be measured in stool samples using immunoassay at baseline and after the intervention (µg/g).

CONTACTS AND LOCATIONS:
Overall Officials: María T Mercader Ros, PhD, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- UCAM San Antonio Catholic University of Murcia, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Abuqwider J, Corrado A, Scida G, Lupoli R, Costabile G, Mauriello G, Bozzetto L. Gut microbiome and blood glucose control in type 1 diabetes: a systematic review. Front Endocrinol (Lausanne). 2023 Nov 15;14:1265696. doi: 10.3389/fendo.2023.1265696. eCollection 2023. PMID 38034007
- [Background] Stewart CJ, Nelson A, Campbell MD, Walker M, Stevenson EJ, Shaw JA, Cummings SP, West DJ. Gut microbiota of Type 1 diabetes patients with good glycaemic control and high physical fitness is similar to people without diabetes: an observational study. Diabet Med. 2017 Jan;34(1):127-134. doi: 10.1111/dme.13140. Epub 2016 May 14. PMID 27100052